CLINICAL TRIAL: NCT01910714
Title: Adapting and Evaluating an Evidence-Based Intervention to Prevent HIV/AIDS Risk Among Apache Youth
Brief Title: Adapting and Evaluating an EBI to Prevent HIV/AIDS Risk Among Apache Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NARCH V: U26IHS300286/03
Record Dates: First submitted 2013-07-17; First posted 2013-07-30 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS; Prevention; American Indian; Substance use; CBPR
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Education Control Condition (Active Comparator): The health education control condition consists of team-building activities and viewing of educational videos on nutrition and fitness, environmental protection and nature. The control condition program will be delivered according to the same structure as the Focus on Youth intervention; daily for 60-90 minutes over the course of 8 days. Due to local staffing availability and the pilot nature of this research, youth in the control condition will not receive the control program in small-group peer format. Rather, youth will receive the control condition program in groups of approximately 30-50.
  Interventions: Behavioral: Health Education Control Condition
- Focus on Youth Intervention (FOY) (Experimental): Focus on Youth is a community-based, eight session group intervention that provides youth with the skills and knowledge they need to protect themselves from HIV and other STDs. Focus on Youth uses fun, interactive activities such as games, role plays and discussions to convey prevention knowledge and skills pertaining to Protection Motivation Theoretical concepts. The intervention consists of 8 group sessions delivered daily over 8 days by two Apache facilitators to same-sex peer groups of 8-12 Apache youth. Each lesson lasts approximately 60-90 minutes. The goal of the sessions will be to teach youth about sexual and reproductive health with a specific focus on safe sex practices and sexual decision making.
  Interventions: Behavioral: Focus On Youth

INTERVENTIONS:
Behavioral: Focus On Youth — Focus on Youth is a community-based, eight session group intervention that provides youth with the skills and knowledge they need to protect themselves from HIV and other STDs. Focus on Youth uses fun, interactive activities such as games, role plays and discussions to convey prevention knowledge and skills pertaining to Protection Motivation Theoretical concepts. The intervention consists of 8 group sessions delivered daily over 8 days by two Apache facilitators to same-sex peer groups of 8-12 Apache youth. Each lesson lasts approximately 60-90 minutes. The goal of the sessions will be to teach youth about sexual and reproductive health with a specific focus on safe sex practices and sexual decision making.
  Arms: Focus on Youth Intervention (FOY)
Behavioral: Health Education Control Condition — The health education control condition consists of team-building activities and viewing of educational videos on nutrition and fitness, environmental protection and nature. The control condition program will be delivered according to the same structure as the Focus on Youth intervention; daily for 60-90 minutes over the course of 8 days. Due to local staffing availability and the pilot nature of this research, youth in the control condition will not receive the control program in small-group peer format. Rather, youth will receive the control condition program in groups of approximately 30-50.
  Arms: Health Education Control Condition

SUMMARY:
The investigators seek to adapt, implement and evaluate a randomized controlled trial of an evidence based intervention delivered by Apache interventionists to reduce HIV/AIDS risk, targeting Apache adolescents. Specific study objectives include:

1. To perform formative research through focus groups and individual interviews on attitudes, practices and intervention preferences among Apache adolescents and community stakeholders.
2. To adapt the Focus on Youth (FOY) evidence-based intervention using findings from the formative research, components of Protection Motivation Theory, and input from a community advisory board.
3. To enroll 304 White Mountain Apache youth ages 13-19 to participate in a randomized intervention trial measuring behavior change at 6- and 12- months follow-up.
4. To determine the feasibility of gathering biological specimens via self-administered swabs to track sexually transmitted diseases among 18-19 year olds enrolled in this and future studies.

DETAILED DESCRIPTION:
The general format of the study consists of a randomized controlled trial delivered through the medium of an 8-day basketball camp. Intervention activities will consist of the daily delivery of a youth HIV/AIDS prevention curriculum over the course of 8 days.

ELIGIBILITY:
Inclusion Criteria:

* American Indian ethnicity and primary residence and/or employment within the White Mountain Apache (Fort Apache) Reservation. Participants must be aged 13-19 years and have parent/guardian consent for youth under 18 years old.

Exclusion Criteria:

* Youth that are unable to fully participate in the evaluation assessments or intervention components will be excluded. In addition, individuals age 16 or older that are listed on either the Federal or Tribal sexual offender registries will be excluded from participation.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 267 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Improved score on condom use self-efficacy scale in treatment vs. control group at 12 months follow-up | 12 months follow-up

SECONDARY OUTCOMES:
Improved score on scale of HIV prevention knowledge, intention and perceptions in treatment vs. control group at 12 months follow-up | 12 months follow-up
Improved score on scale of partner negotiation skills related to sex and drug use between treatment vs. control group at 12 months follow-up | 12 months follow-up
Higher use of condoms at last sex in treatment vs. control group at 12 months follow-up | 12 months follow-up
Less frequency of sex with substance use in treatment vs. control group at 12 months follow-up | 12 months follow-up
Higher age of sexual initiation in treatment vs. control group at 12 months follow-up | 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Anne Rompalo, MD, ScM, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Center for American Indian Health, Baltimore, Maryland, United States